CLINICAL TRIAL: NCT02781922
Title: Efficacy and Safety Study of Autologous Cardiac Stem Cells (JRM-001) Treated After Reconstructive Surgery in Pediatric Patients With Congenital Heart Disease: A Multicenter Randomized Single-blind Parallel-group Study
Brief Title: Cardiac Stem/Progenitor Cell Infusion in Univentricular Physiology (APOLLON Trial)
Acronym: APOLLON
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Metcela Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001-CLJ-001
Record Dates: First submitted 2016-05-19; First posted 2016-05-25 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: Hypoplastic Left Heart Syndrome; Single Ventricle
Keywords: cardiac stem/progenitor cells; autologous cell therapy; functional single ventricle; congenital heart disease
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Univentricular Heart; Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autologous cardiac stem cells (JRM-001) (Experimental)
  Interventions: Genetic: Autologous cardiac stem cells (JRM-001)
- Usual care (No Intervention)

INTERVENTIONS:
Genetic: Autologous cardiac stem cells (JRM-001) — 3x 10^5 cells/kg, single treatment
  Arms: Autologous cardiac stem cells (JRM-001)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of intracoronary injection of JRM-001 after reconstructive surgery in pediatric patients with functional single ventricle

ELIGIBILITY:
Inclusion Criteria:

* Functional single ventricle patient with heart failure who is scheduled for stage 2 (Glenn) or stage 3 (Fontan) surgery
* EF(%) by echocardiography ≤ 55%
* Able to obtain written informed consent of participation in the study by a parent of the patient

Exclusion Criteria:

* Known medical history of cardiogenic shock
* Lethal, uncontrollable arrhythmia
* Complication of coronary artery disease
* Eisenmenger syndrome
* Complication of brain dysfunction due to circulatory failure
* Malignant neoplasm
* Complication of severe neurologic disorder
* Severe pulmonary embolism or pulmonary hypertension
* Severe renal failure
* Multiple organ failure
* Active infection (including endocarditis)
* Sepsis
* Active hemorrhagic disease (e.g. gastrointestinal bleeding, injury)
* Known history of hypersensitivity to anti-infective drugs
* Inability to complete the protocol treatment and baseline to follow-up examinations

Ages: 0 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in ejection fraction (EF(%)) assessed by MRI from baseline | Baseline, 6 and 12 months

SECONDARY OUTCOMES:
Change in EF(%) assessed by echocardiograms from baseline | Screening, Baseline, 3, 6 and 12 months
Change in EF(%) assessed by cardiac catheterization from baseline | Baseline, 6 and 12 months
Change in Ea/Ees assessed by cardiac catheterization from baseline | Baseline, 6 and 12 months
Change in Ventricular Stiffness assessed by cardiac catheterization from baseline | Baseline, 6 and 12 months
Change in heart failure index from baseline | Baseline, 3, 6 and 12 months
Change in Quality of Life (QOL) index from baseline | Baseline, 6 and 12 months
Number of adverse events | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (4):
  - Kanagawa Children's Medical Center, Kanagawa
  - Okayama University Hospital, Okayama
  - Saitama Prefectural Children's Medical Center, Saitama
  - Shizuoka Children's Hospital, Shizuoka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishigami S, Ohtsuki S, Tarui S, Ousaka D, Eitoku T, Kondo M, Okuyama M, Kobayashi J, Baba K, Arai S, Kawabata T, Yoshizumi K, Tateishi A, Kuroko Y, Iwasaki T, Sato S, Kasahara S, Sano S, Oh H. Intracoronary autologous cardiac progenitor cell transfer in patients with hypoplastic left heart syndrome: the TICAP prospective phase 1 controlled trial. Circ Res. 2015 Feb 13;116(4):653-64. doi: 10.1161/CIRCRESAHA.116.304671. Epub 2014 Nov 17. PMID 25403163
- [Background] Tarui S, Ishigami S, Ousaka D, Kasahara S, Ohtsuki S, Sano S, Oh H. Transcoronary infusion of cardiac progenitor cells in hypoplastic left heart syndrome: Three-year follow-up of the Transcoronary Infusion of Cardiac Progenitor Cells in Patients With Single-Ventricle Physiology (TICAP) trial. J Thorac Cardiovasc Surg. 2015 Nov;150(5):1198-1207, 1208.e1-2. doi: 10.1016/j.jtcvs.2015.06.076. Epub 2015 Jul 8. PMID 26232942
- [Background] Ishigami S, Ohtsuki S, Eitoku T, Ousaka D, Kondo M, Kurita Y, Hirai K, Fukushima Y, Baba K, Goto T, Horio N, Kobayashi J, Kuroko Y, Kotani Y, Arai S, Iwasaki T, Sato S, Kasahara S, Sano S, Oh H. Intracoronary Cardiac Progenitor Cells in Single Ventricle Physiology: The PERSEUS (Cardiac Progenitor Cell Infusion to Treat Univentricular Heart Disease) Randomized Phase 2 Trial. Circ Res. 2017 Mar 31;120(7):1162-1173. doi: 10.1161/CIRCRESAHA.116.310253. Epub 2017 Jan 4. PMID 28052915